CLINICAL TRIAL: NCT05878574
Title: Prospective Cohort Study of Bone Mineral Density and Calcium-phosphorus Metabolism in RSA Patients: Low Molecular Weight Heparin Use Versus Control
Brief Title: Prospective Study of BMD and Ca-P Metabolism in RSA Patients: LMWH Use Versus Control
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aimin Zhao (Other)
Responsible Party: Sponsor-Investigator, Aimin Zhao, Director of Obstetrics and Gynecology, RenJi Hospital
Organization: RenJi Hospital (Other)
Other Study IDs: IIT-2023-0010
Record Dates: First submitted 2023-05-07; First posted 2023-05-26 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Recurrent Spontaneous Abortion
MeSH Terms: conditions — Abortion, Spontaneous | interventions — Heparin, Low-Molecular-Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LMWH group: Continuous use of low molecular weight heparin for more than 3 months during pregnancy preparation and during pregnancy with a history of more than 2 consecutive miscarriages before 28 weeks of gestation
  Interventions: Drug: Low molecular weight heparin
- control group: No use of low molecular weight heparin during pregnancy preparation and throughout pregnancy and history of more than 2 consecutive miscarriages before 28 weeks of gestation

INTERVENTIONS:
Drug: Low molecular weight heparin — Continuous use of LMWH for more than 3 months during pregnancy preparation and through pregnancy
  Other Names: LMWH
  Groups: LMWH group

SUMMARY:
The goal of this prospective observational study is to learn about the effect of low molecular weight heparin (LMWH) application on bone mineral density (BMD) and on calcium-phosphorus metabolism in patients with recurrent spontaneous abortion (RSA), and to compare the degree of bone loss and changes in blood calcium and phosphorus in RSA patients and in control groups with normal pregnancy. By monitoring ultrasound BMD and serum indicators related to maternal bone formation and Ca-P metabolism, the association mechanism between long-term use of LMWH, maternal Ca-P regulation and bone loss will be constructed, so as to contribute to clinical treatment and lifestyle guidance during pregnancy in RSA patients.

DETAILED DESCRIPTION:
Women who meet the inclusion criteria at the outpatient clinic of Renji Hospital are recruited in this study from November 2022 to December 2023. Basic information of all subjects is recorded, including number of miscarriages, duration of breastfeeding, comorbidities, and intake of nutritional supplements. Subjects' medication use during the study is recorded as well. Subjects will undergo ultrasound BMD at six time points: before and after medication during pregnancy preparation, at 10, 24, 32 weeks of pregnancy, and at 42 days postpartum. Peripheral blood will also be collected at the time points above to measure serum osteocalcin, blood calcium, blood phosphorus, 25(OH) D, thyroid hormone, and parathyroid hormone levels. Subjects will be followed up to 42 days postpartum to observe pregnancy outcomes and health conditions of the newborn.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 45 years.
* Female who needs to prepare for pregnancy or have a confirmed pregnancy
* normal karyotype of chromosomes.
* normal uterine anatomy under pelvic ultrasound examination.
* Cooperation in completing blood sample collection, testing and ultrasound examination.
* no serious medical or surgical comorbidities.
* Sign the informed consent form.

Exclusion Criteria:

* Presence of diseases affecting calcium metabolism, including primary hyperparathyroidism, Cushing's disease, chronic liver, kidney and gastrointestinal (e.g., celiac disease) disorders and rheumatoid arthritis.
* Known HIV positive and / or screening visit, HBsAg or HCV antibody positive.
* The malignant tumors occurred in the past 5 years (except for the skin squamous basal cell carcinoma which has been resected and considered cured). Subjects who developed malignancies five years ago should provide evidence of remission or cure. Subjects with a history of cervical cancer who had undergone conization or cure in the past 3 years were eligible.
* Patients with a history of chronic infection such as Mycoplasma, chlamydia, Cryptococcus and invasive fungal infection should be discussed with the main researchers.
* History of active tuberculosis (TB) or evidence of previous TB infection. Subjects with a history of potential TB infection should also be excluded, unless there is a documented evidence that they have completed appropriate anti TB treatment in accordance with CDC guidelines or local regulations before screening. In addition, subjects were strictly forbidden to have any clinical symptoms / signs of active TB.
* Presence of pregnancy contraindications.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All women with a need for pregnancy preparation or a confirmed pregnancy who meet the inclusion criteria from November 2022 to December 2023 at the outpatient clinic of Renji Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 344 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
ultrasound BMD before medication during pregnancy preparation | 4 weeks
  use ultrasound to test heel bone mineral density before medication during pregnancy preparation
ultrasound BMD after medication during pregnancy preparation | up to 16 weeks
  use ultrasound to test heel bone mineral density after medication during pregnancy preparation
ultrasound BMD at 10th weeks of pregnancy | up to 26 weeks
  use ultrasound to test heel bone mineral density at 10th weeks of pregnancy
ultrasound BMD at 24th weeks of pregnancy | 40 weeks
  use ultrasound to test heel bone mineral density at 24th weeks of pregnancy
ultrasound BMD at 32nd weeks of pregnancy | 1 year
  use ultrasound to test heel bone mineral density at 32nd weeks of pregnancy
ultrasound BMD at postpartum | up to 1 year and 2 months
  use ultrasound to test heel bone mineral density at postpartum

SECONDARY OUTCOMES:
osteocalcin before medication during pregnancy preparation | 4 weeks
  use peripheral blood test to detect N-terminal mid-molecular fragment of serum osteocalcin before medication during pregnancy preparation
osteocalcin after medication during pregnancy preparation | up to 16 weeks
  use peripheral blood test to detect N-terminal mid-molecular fragment of serum osteocalcin after medication during pregnancy preparation
osteocalcin at 10th weeks of pregnancy | up to 26 weeks
  use peripheral blood test to detect N-terminal mid-molecular fragment of serum osteocalcin at 10th weeks of pregnancy
osteocalcin at 24th weeks of pregnancy | 40 weeks
  use peripheral blood test to detect N-terminal mid-molecular fragment of serum osteocalcin at 24th weeks of pregnancy
osteocalcin at 32nd weeks of pregnancy | 1 year
  use peripheral blood test to detect N-terminal mid-molecular fragment of serum osteocalcin at 32nd weeks of pregnancy
osteocalcin at postpartum | up to 1 year and 2 months
  use peripheral blood test to detect N-terminal mid-molecular fragment of serum osteocalcin at postpartum
calcium before medication during pregnancy preparation | 4 weeks
  use peripheral blood test to detect calcium level before medication during pregnancy preparation
calcium after medication during pregnancy preparation | up to 16 weeks
  use peripheral blood test to detect calcium level after medication during pregnancy preparation
calcium at 10th weeks of pregnancy | up to 26 weeks
  use peripheral blood test to detect calcium level at 10th weeks of pregnancy
calcium at 24th weeks of pregnancy | 40 weeks
  use peripheral blood test to detect calcium level at 24th weeks of pregnancy
calcium at 32nd weeks of pregnancy | 1 year
  use peripheral blood test to detect calcium level at 32nd weeks of pregnancy
calcium at postpartum | up to 1 year and 2 months
  use peripheral blood test to detect calcium level at postpartum
PTH before medication during pregnancy preparation | 4 weeks
  use peripheral blood test to detect parathyroid hormone level before medication during pregnancy preparation
PTH after medication during pregnancy preparation | up to 16 weeks
  use peripheral blood test to detect parathyroid hormone level after medication during pregnancy preparation
PTH at 10th weeks of pregnancy | up to 26 weeks
  use peripheral blood test to detect parathyroid hormone level at 10th weeks of pregnancy
PTH at 24th weeks of pregnancy | 40 weeks
  use peripheral blood test to detect parathyroid hormone level at 24th weeks of pregnancy
PTH at 32nd weeks of pregnancy | 1 year
  use peripheral blood test to detect parathyroid hormone level at 32nd weeks of pregnancy
PTH at postpartum | up to 1 year and 2 months
  use peripheral blood test to detect parathyroid hormone level at postpartum
live bitrh | 1 year
  A live baby born after 23 weeks of gestation

CONTACTS AND LOCATIONS:
Overall Officials: Aimin Zhao, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No